CLINICAL TRIAL: NCT03201211
Title: A Long-term Follow-up Study of the Investigational GSK Biologicals' GSK3277511A Vaccine in Adults
Brief Title: A Long Term Follow-up Study up to 4 Years After Study Vaccination to Assess Immunogenicity and Safety of the Investigational Vaccine in Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 204913; 2016-004248-13 (EudraCT Number)
Record Dates: First submitted 2017-06-19; First posted 2017-06-28 (Actual); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Respiratory Disorders
Keywords: Safety; Immunogenicity
MeSH Terms: conditions — Respiration Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 10-10-10-AS (Experimental): Subjects who received two doses of the AS01E adjuvanted GSK Biologicals' NTHi-Mcat investigational vaccine, containing 10µg of PD, PE-PilA and UspA2, and administered at Month 0 and Month 2 in NTHi-Mcat-001 study (NCT02547974), and were enrolled in the study.
  Interventions: Biological: Blood sampling; Biological: GSK biologicals investigational NTHi Mcat vaccine containing 10µg of PD, PE-PilA and UspA2.
- 10-10-3-AS (Experimental): Subjects who received two doses of the AS01E adjuvanted GSK Biologicals' NTHi-Mcat investigational vaccine, containing 10µg of PD, 10µg of PE-PilA, and 3.3µg of UspA2, and administered at Month 0 and Month 2 in NTHi-Mcat-001 study (NCT02547974), and were enrolled in the study.
  Interventions: Biological: Blood sampling; Biological: GSK biologicals investigational NTHi Mcat vaccine containing 10µg of PD, 10µg of PE-PilA, and 3.3µg of UspA2.
- PLACEBO (Placebo Comparator): Subjects who received two doses of placebo (saline solution), administered at Month 0 and Month 2 in NTHi-Mcat-001 study (NCT02547974) and were enrolled in the study.
  Interventions: Biological: Blood sampling; Drug: Placebo

INTERVENTIONS:
Biological: Blood sampling — A volume of approximately 20 mL of whole blood should be drawn from each subject, at each study visit, for antibody determination and assay validation/development.
Biological: GSK biologicals investigational NTHi Mcat vaccine containing 10µg of PD, PE-PilA and UspA2. — 2 doses, not administered as part of this study but administered at Day 0 and Day 60 during STEP 2 of NTHi Mcat-001 (201281 - NCT02547974) study, to subjects who were then enrolled in this study. Intramuscular vaccination in the deltoid region of the non-dominant arm according to protocol schedule.
  Arms: 10-10-10-AS
Biological: GSK biologicals investigational NTHi Mcat vaccine containing 10µg of PD, 10µg of PE-PilA, and 3.3µg of UspA2. — 2 doses, not administered as part of this study but administered at Day 0 and Day 60 during STEP 2 of NTHi Mcat-001 (201281 - NCT02547974) study, to subjects who were then enrolled in this study. Intramuscular vaccination in the deltoid region of the non-dominant arm according to protocol schedule.
  Arms: 10-10-3-AS
Drug: Placebo — 2 doses, not administered as part of this study but administered at Day 0 and Day 60 during STEP 2 of NTHi Mcat-001 (201281 - NCT02547974) study, to subjects who were then enrolled in this study. Intramuscular vaccination in the deltoid region of the non-dominant arm according to protocol schedule.
  Arms: PLACEBO

SUMMARY:
The purpose of this long-term follow-up of a Phase I study is to evaluate the kinetics of the antibody response to NTHi-Mcat antigens and long-term safety, in subjects aged between 50-71 years at the time of enrolment in the NTHi-Mcat-001 study. These subjects were previously exposed to two adjuvanted formulations of the NTHi-Mcat vaccine administered according to a 0, 2 months schedule in the NTHi-Mcat-001 (201281) study. The subjects that had received saline placebo controls will also be included in this follow-up study to make comparisons with the investigational vaccines. No vaccinations will be administered in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who previously participated in STEP 2 of study NTHi-Mcat-001 (201281), and performed the last study visit (Month 14) and received the 2 study vaccinations.
* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g. return for follow-up visits). And subjects' Legally Acceptable Representative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply, with the requirements of the protocol.
* Written informed consent obtained from the subject/ LAR(s) of the subject prior to performance of any study specific procedure.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) during the period starting 30 days before the first follow-up study visit (Month 19 to Month 20), or planned use during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs since the end of the NTHi-Mcat-001 study. For corticosteroids, this will mean prednisone ≥ 20 mg/day, or equivalent. Inhaled and topical steroids are allowed.
* Administration of long-acting immune-modifying drugs at any time during the study period (e.g. infliximab).
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device).
* Administration of immunoglobulins and/or any blood products during the period starting 3 months before the first follow-up visit or planned administration during the study period.
* Current alcoholism and/or drug abuse.
* Has significant disease (including significant neurological or psychological disorders), in the opinion of the investigator, likely to interfere with the study and/or likely to cause death within the study duration.
* Any other condition that the investigator judges may interfere with study findings.

Ages: 51 Years to 73 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Belgium (3):
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Wilrijk

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Groups:
- 10-10-3-AS: Subjects who received two doses of the AS01E-adjuvanted GSK Biologicals' NTHi-Mcat investigational vaccine, containing 10µg of PD, 10µg of PE-PilA, and 3.3µg of UspA2, and administered at Month 0 and Month 2 in NTHi-Mcat-001 study (NCT02547974), and were enrolled in the study.
Period: Overall Study
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Started | 27 | 26 | 28
Completed | 25 | 25 | 27
Not Completed | 2 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — CONSENT WITHDRAWAL NOT DUE TO ADV. EVENT | 0 | 0 | 1
Not completed — OTHER unknown reasons | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO | Total
Number analyzed (Participants) | 27 | 26 | 28 | 81
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.7 (6.3) | 59.0 (5.9) | 58.2 (6.5) | 58.9 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 9 | 33
  Male | 15 | 14 | 19 | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  WHITE - CAUCASIAN / EUROPEAN HERITAGE | 27 | 26 | 28 | 81

OUTCOME MEASURES:

1. Primary Outcome: Anti-Protein D (PD) Antibody Concentrations, Measured as Component of the NTHi Mcat Investigational Vaccine
Description: Adjusted geometric mean concentration (GMC) and their 95% confidence interval (CI) was calculated. GMCs were estimated using an ANCOVA model including treatment group as fixed effect and Month 0 antibody concentration from NTHi Mcat-001 as covariate. The cut-off value of the enzyme-linked immunosorbent assay (ELISA) anti-PD assay was 153 ELISA unit per millilitre (EU/mL).
Time Frame: At Month 20
Population: Analysis was performed on the Per Protocol Set (PPS) which included all subjects enrolled in this study, who provided informed consent, complied with the eligibility criteria, study procedures and with immunogenicity data for specified antibody at specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 26 | 26 | 28
EU/mL | 382.7 [279.2 to 524.4] | 511.9 [376.4 to 696.2] | 90.5 [67.1 to 121.9]

2. Primary Outcome: Anti-PD Antibody Concentrations, Measured as Component of the NTHi Mcat Investigational Vaccine
Description: Adjusted GMC and their 95% CI was calculated. GMCs were estimated using an ANCOVA model including treatment group as fixed effect and Month 0 antibody concentration from NTHi Mcat-001 as covariate. The cut-off value of the ELISA anti-PD assay was 153 EU/mL.
Time Frame: At Month 26
Population: Analysis was performed on the PPS which included all subjects enrolled in this study, who provided informed consent, complied with the eligibility criteria, study procedures and with immunogenicity data for specified antibody at specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 26 | 26 | 27
EU/mL | 373.4 [270.2 to 516.1] | 537.2 [392.8 to 734.7] | 93.2 [68.4 to 127.0]

3. Primary Outcome: Anti-PD Antibody Concentrations, Measured as Component of the NTHi Mcat Investigational Vaccine
Description: as for outcome 2
Time Frame: At Month 32
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 25 | 26 | 27
EU/mL | 371.8 [271.4 to 509.5] | 480.8 [356.2 to 649.0] | 94.1 [70.0 to 126.6]

4. Primary Outcome: Anti-PD Antibody Concentrations, Measured as Component of the NTHi Mcat Investigational Vaccine
Description: as for outcome 2
Time Frame: At Month 38
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 24 | 26 | 27
EU/mL | 368 [264.4 to 512.0] | 490.4 [358.0 to 671.8] | 99.8 [73.1 to 136.2]

5. Primary Outcome: Anti-PD Antibody Concentrations, Measured as Component of the NTHi Mcat Investigational Vaccine
Description: as for outcome 2
Time Frame: At Month 44
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 25 | 26 | 27
EU/mL | 321.4 [235.1 to 439.2] | 466.2 [346.4 to 627.6] | 95.6 [71.2 to 128.3]

6. Primary Outcome: Anti-PD Antibody Concentrations, Measured as Component of the NTHi Mcat Investigational Vaccine
Description: as for outcome 2
Time Frame: At Month 50
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 25 | 23 | 27
EU/mL | 315.4 [225.5 to 441.1] | 474.5 [337.9 to 666.3] | 101.5 [74.0 to 139.3]

7. Primary Outcome: Anti-Protein E (PE) Antibody Concentrations, Measured as Component of the NTHi Mcat Investigational Vaccine
Description: Adjusted GMC and their 95% CI was calculated. GMCs were estimated using an ANCOVA model including treatment group as fixed effect and Month 0 antibody concentration from NTHi Mcat-001 as covariate. The cut-off value of the ELISA anti-PE assay was 8 EU/mL.
Time Frame: At Month 20
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 27 | 26 | 28
EU/mL | 762.7 [549.4 to 1058.6] | 1215 [869.5 to 1697.9] | 21.5 [15.6 to 29.6]

8. Primary Outcome: Anti-PE Antibody Concentrations, Measured as Component of the NTHi Mcat Investigational Vaccine
Description: as for outcome 7
Time Frame: At Month 26
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 26 | 26 | 27
EU/mL | 729.5 [519.2 to 1024.9] | 1258.9 [895.5 to 1769.9] | 23.1 [16.6 to 32.3]

9. Primary Outcome: Anti-PE Antibody Concentrations, Measured as Component of the NTHi Mcat Investigational Vaccine
Description: as for outcome 7
Time Frame: At Month 32
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 25 | 26 | 27
EU/mL | 603.9 [424.1 to 859.8] | 998.1 [705.4 to 1412.2] | 19.3 [13.7 to 27.1]

10. Primary Outcome: Anti-PE Antibody Concentrations, Measured as Component of the NTHi Mcat Investigational Vaccine
Description: Adjusted GMC and their 95% CI was calculated. GMCs were estimated using an ANCOVA model including treatment group as fixed effect and Month 0 antibody concentration from NTHi Mcat-001 as covariate. The cut-off value of the F13ELISA anti-PE assay was 8 EU/mL.
Time Frame: At Month 38
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 24 | 26 | 27
EU/mL | 596 [414.8 to 856.4] | 1003.7 [708.0 to 1422.8] | 20.2 [14.4 to 28.5]

11. Primary Outcome: Anti-PE Antibody Concentrations, Measured as Component of the NTHi Mcat Investigational Vaccine
Description: as for outcome 7
Time Frame: At Month 44
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 25 | 26 | 27
EU/mL | 524.8 [373.4 to 737.6] | 782.6 [560.5 to 1092.9] | 19.4 [14.0 to 27.0]

12. Primary Outcome: Anti-PE Antibody Concentrations, Measured as Component of the NTHi Mcat Investigational Vaccine
Description: as for outcome 7
Time Frame: At Month 50
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 25 | 23 | 27
EU/mL | 491.3 [342.5 to 704.5] | 827.8 [568.3 to 1205.7] | 22 [15.6 to 31.2]

13. Primary Outcome: Anti-type IV Pili Subunit (PilA) Antibody Concentrations, Measured as Component of the NTHi Mcat Investigational Vaccine
Description: Adjusted GMC and their 95% CI was calculated. GMCs were estimated using an ANCOVA model including treatment group as fixed effect and Month 0 antibody concentration from NTHi Mcat-001 as covariate.The cut-off value of the ELISA anti-PilA assay was 7 EU/mL.
Time Frame: At Month 20
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 27 | 26 | 28
EU/mL | 121.9 [91.0 to 163.4] | 188.3 [139.5 to 254.2] | 13.8 [10.3 to 18.6]

14. Primary Outcome: Anti-PilA Antibody Concentrations, Measured as Component of the NTHi Mcat Investigational Vaccine
Description: as for outcome 13
Time Frame: At Month 26
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 26 | 26 | 27
EU/mL | 96.4 [73.2 to 126.9] | 171.6 [130.1 to 226.4] | 13 [9.9 to 17.2]

15. Primary Outcome: Anti-PilA Antibody Concentrations, Measured as Component of the NTHi Mcat Investigational Vaccine
Description: as for outcome 13
Time Frame: At Month 32
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 25 | 26 | 27
EU/mL | 79.7 [57.5 to 110.5] | 166.9 [121.0 to 230.3] | 10 [7.2 to 13.8]

16. Primary Outcome: Anti-PilA Antibody Concentrations, Measured as Component of the NTHi Mcat Investigational Vaccine
Description: as for outcome 13
Time Frame: At Month 38
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 24 | 26 | 27
EU/mL | 68 [48.6 to 95.2] | 147.5 [106.6 to 204.2] | 9.6 [6.9 to 13.3]

17. Primary Outcome: Anti-PilA Antibody Concentrations, Measured as Component of the NTHi Mcat Investigational Vaccine
Description: as for outcome 13
Time Frame: At Month 44
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 25 | 26 | 27
EU/mL | 60.8 [44.4 to 83.3] | 122.5 [89.8 to 167.0] | 10.2 [7.5 to 13.9]

18. Primary Outcome: Anti-PilA Antibody Concentrations, Measured as Component of the NTHi Mcat Investigational Vaccine
Description: as for outcome 13
Time Frame: At Month 50
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 25 | 23 | 27
EU/mL | 54.2 [39.0 to 75.3] | 106.5 [75.6 to 150.1] | 9.8 [7.1 to 13.6]

19. Primary Outcome: Anti-ubiquitous Surface Protein A2 of Moraxella Catarrhalis (UspA2) Antibody Concentrations, Measured as Component of the NTHi Mcat Investigational Vaccine
Description: Adjusted GMC and their 95% CI was calculated. GMCs were estimated using an ANCOVA model including treatment group as fixed effect and Month 0 antibody concentration from NTHi Mcat-001 as covariate.The cut-off value of the ELISA anti-UspA2 assay was 18 EU/mL.
Time Frame: At Month 20
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 27 | 26 | 28
EU/mL | 719 [600.9 to 860.2] | 578.2 [481.5 to 694.3] | 456.1 [382.7 to 543.6]

20. Primary Outcome: Anti-UspA2 Antibody Concentrations, Measured as Component of the NTHi Mcat Investigational Vaccine
Description: as for outcome 19
Time Frame: At Month 26
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 26 | 26 | 27
EU/mL | 791.1 [638.0 to 981.0] | 621.6 [501.4 to 770.6] | 480.4 [389.5 to 592.7]

21. Primary Outcome: Anti-UspA2 Antibody Concentrations, Measured as Component of the NTHi Mcat Investigational Vaccine
Description: as for outcome 19
Time Frame: At Month 32
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 25 | 26 | 26
EU/mL | 666.6 [556.9 to 797.8] | 530.5 [444.7 to 632.8] | 434.7 [364.8 to 517.9]

22. Primary Outcome: Anti-UspA2 Antibody Concentrations, Measured as Component of the NTHi Mcat Investigational Vaccine
Description: as for outcome 19
Time Frame: At Month 38
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 24 | 26 | 27
EU/mL | 662.3 [531.8 to 824.8] | 556.6 [451.2 to 686.7] | 453.2 [369.2 to 556.3]

23. Primary Outcome: Anti-UspA2 Antibody Concentrations, Measured as Component of the NTHi Mcat Investigational Vaccine
Description: as for outcome 19
Time Frame: At Month 44
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 25 | 26 | 27
EU/mL | 561.5 [451.9 to 697.6] | 400.1 [323.3 to 495.2] | 339.4 [275.7 to 417.8]

24. Primary Outcome: Anti-UspA2 Antibody Concentrations, Measured as Component of the NTHi Mcat Investigational Vaccine
Description: as for outcome 19
Time Frame: At Month 50
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 25 | 23 | 27
EU/mL | 536.8 [424.0 to 679.6] | 404.5 [316.0 to 517.7] | 374.9 [299.2 to 469.8]

25. Secondary Outcome: Number of Subjects Reported With Any Serious Adverse Event (SAE)
Description: A SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalisation or prolongation of existing hospitalisation, results in disability/incapacity.
Time Frame: From first visit (Month 20) up to study conclusion (Month 50)
Population: Analysis was performed on all the subjects enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 27 | 26 | 28
Participants | 5 | 2 | 2

26. Secondary Outcome: Number of Subjects Reported With Any Potential Immune-mediated Disease (pIMD)
Description: pIMD's are a subset of Adverse Events that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: From first visit (Month 20) up to study conclusion (Month 50)
Population: Analysis was performed on all the subjects enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
Number analyzed (Participants) | 27 | 26 | 28
Participants | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: SAEs were collected from first visit (Month 20) up to study conclusion (Month 50). Other adverse events were not collected during the study period.
Description: Other AEs are not collected in the study as no administration of vaccine.
Arm/Group | 10-10-10-AS | 10-10-3-AS | PLACEBO
All-Cause Mortality (participants affected / at risk) | 1/27 | 0/26 | 0/28
Serious Adverse Events (participants affected / at risk) | 5/27 | 2/26 | 2/28
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10-10-10-AS (N=27) | 10-10-3-AS (N=26) | PLACEBO (N=28)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT03201211/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/11/NCT03201211/SAP_001.pdf